CLINICAL TRIAL: NCT06646471
Title: PROspective Master-protocol for Evaluation of Systemic THErapeutics in Elderly
Brief Title: PROspective Master-protocol for Evaluation of Systemic THErapeutics in Elderly With Thoracic Malignancies
Acronym: PROMETHEE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: GFPC Investigation (Other)
Responsible Party: Sponsor
Organization: Groupe Francais De Pneumo-Cancerologie (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GFPC 05-2023
Record Dates: First submitted 2024-09-27; First posted 2024-10-17 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-08

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Real world cohort of NSCLC older adults patients (Other): Cohort of patients ≥70 years of age with NSCLC treated in first line therapy for thoracic tumors according to ESMO-referenced therapeutic standards or according to an innovative molecule and/or strategy.
  An optional biobank based on blood samples taken during the screening phase prior to the first administration of systemic treatment will be collected. Sampling of tumoral materials will be collected prior to study participation and send for central reading.
  Patients will be asked to come at the hospital for their regular visits as per site current practice and to complete three quality of life questionnaires (EORTC QLQ-F17; QLQ-LC13; QLQ-ELD14).
  Interventions: Genetic: Bio-bank repository; Other: Quality of Life (QoL); Procedure: G-Code

INTERVENTIONS:
Genetic: Bio-bank repository — Blood samples taken during the screening phase prior to the first administration of systemic treatment and stored in a repository for a maximum duration of 10 years
Other: Quality of Life (QoL) — Collection of EORTC QoL questionnaires QLQ-F17, QLQ-LC13 and QLQ-ELD14:
  * stage 3 non-operable/non-radiable, stage 4: at inclusion, 12 weeks, 6 months of treatment, first-line progression.
  * operable stage 1 to 3b: at inclusion, end of neoadjuvant period before surgery post-operative baseline, at 6 months, at 12 months.
  * radiable stages 3a to 3c: at inclusion, at the end of thoracic radiotherapy, at 6 months, at 12 months.
Procedure: G-Code — G-CODE: Katz Autonomy Scale (ADL), Instrumental Activities of Daily Living questionnaire (IADL), Charlson score, mini GDS, mini COG, falls history, Timed Get Up and Go test, social environment.

SUMMARY:
The objective of the study is to prospectively generate real-life data in patients aged ≥70 years treated in first line for a thoracic tumor (Non-Small-Cell Lung Carcinoma) according to best standard of care as defined by the European Society for Medical Oncology (ESMO). This cohort will aim to:

* characterize participants in terms of geriatrics, biology and carcinology
* describe the treatment modalities by stage, as well as the results in terms of efficacy, safety and impact on quality of life.

At the same time, exploratory sub-cohorts will be identified including participants treated uniformly with the same molecule, and/or the same innovative strategy.

Participants will be followed in accordance with investigator's usual clinical practice at the corresponding site. They will be asked to:

* visit the clinic as per physician's request for checkups and tests for assessing general condition and clinical efficacy and tolerance of current treatment.
* perform the necessary regular para-clinical examinations (lab testing, imaging, re-biopsy).
* provide blood samples for bio-bank repository
* perform assessments specific to older adults
* answer three quality of life questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥70 years
* Non-small-cell lung cancer for which the multidisciplinary consultation required systemic treatment regardless of Tumor-Node-Metastasis (TNM) stage
* Patient naïve to systemic anticancer treatment for bronchial neoplasia
* Patient covered by social security
* Patient eligible for systemic treatment
* Systemic treatment with marketing authorization in the indication, available in routine care early access or compassionate access.
* Patient able to understand the protocol
* Patient not opposed to the collection of data concerning him/her
* Signature of study consent form.

Exclusion Criteria:

* Patients under guardians or curators
* Patient not under the care of the investigating center and not monitored by the investigating center
* Patient already treated with systemic therapy for NSCLC

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From the date of first dose of treatment received until the date of the first documented disease progression according to Response Evaluation Criteria in Solid Tumor (RECIST) 1.1 or to death from any cause, whichever comes first, assessed up to 2 years
  The Progression Free Survival is defined as the time between treatment start date and event date defined by the Response Evaluation Criteria in Solid Tumor (RECIST) 1.1 progression or death for any cause, whichever comes first.
  Disease progression will be evaluated according to (RECIST) 1.1 assessed locally. Frequency of this assessment is let to the investigator 's discretion and local practices.
  The participants will be followed until disease progression or death for any cause. Patients without an event at the time of analysis will be censored at the date of their last tumor assessment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From the date of first dose of treatment received until the date of the first documented disease progression according to Response Evaluation Criteria in Solid Tumor (RECIST) 1.1 or to death from any cause, whichever comes first, assessed up to 2 years
  The objective response rate (ORR) is defined as the proportion of patients with complete response (CR) or partial response (PR) as the best response during the study according to RECIST 1.1 criteria based on tumoral assessment performed by thorax-abdominal-pelvic and brain CT scans. The frequency of the tumor assessments will follow the site practices.
Overall Survival (OS) | From the treatment start date up to the date of death for a 2-year-period maximum
  Overall survival (OS) is calculated as the time between the date of treatment initiation and date of death, and censored at date of last news for patients alive at the end of the study.
Duration of Response (DOR) | From the date of the first response to the date of progression or death, whichever comes first, or for a 2-year-period maximum
  The duration of response is defined as the time between the date of the first response assessed by RECIST 1.1 to the date of progression or death for any cause, whichever comes first, and censored at the date of last tumor evaluation for patients still responding to treatment at the end of the study (after 2 years).
Time to Response (TTR) | From the start date of treatment up to the date of first response or for a 2-year-period maximum
  Time to response is measured from the date of treatment initiation to the date of first response as defined by RECIST 1.1.
Treatment Duration | From the treatment start date and the treatment stop date whatever the cause up to a 2-year-period maximum.
  The duration of treatment is defined as the time between the treatment start date and the date of definitive cessation of treatment, whatever the cause.
Safety events | From the enrollment up to the participants study end date or for a 2-year-period maximum
  All adverse events experienced by the participants, whatever the grades of toxicity, will be collected according to CTCAE v4.0 (common terminology criteria for adverse events).
Treatments description | From the start date of the NSCLC treatment up to the participant study end date or for a 2-year-period maximum
  The treatments for NSCLC will be described including the adaptations: discontinuations, treatment interruptions, dose adaptations. The reasons for the changes will be recorded.
Geriatric interventions: specialized consultations | From the enrollment up to the participant study end date or for a 2-year-period maximum
  The specialized geriatric consultations carried out to correct frailties will be collected during the study participation including psychological and/or dietetic consultations.
Geriatric interventions: specialized exercises | From the enrollment up to the participant study end date or for a 2-year-period maximum
  The specialized geriatric exercises carried out to correct frailties will be collected during the study participation including prescription of adapted physical activity and/or cognitive stimulation exercises.
Geriatric interventions: specialized help at home | From the enrollment up to the participant study end date or for a 2-year-period maximum
  The specialized geriatric interventions at home carried out to correct frailties will be collected during the study participation including home visits by a nurse or home help.
Geriatric interventions: specialized medications | From the enrollment up to the participant study end date or for a 2-year-period maximum
  The specialized geriatric medications carried out to correct frailties will be collected during the study participation.
European Organisation for Research and Treatment of Cancer Core Function Questionnaire (QLQ-F17) | At enrolment, at 12 weeks, at 6 months and at 12 months.
  The QLQ-F17 is a validated cancer-specific questionnaire specific to cancer. It includes 17 items to assess 6 QoL scales: 1 global health scale and 5 functional scales (physical, role,emotional, cognitive, social). This is a shortened version of the QLQ-C30, containing only the functional and overall quality of life sections. This questionnaire was developed by the EORTC in order to optimize the collection of quality-of-life data, and to avoid overloading the patient with a lengthy questionnaire.
  Symptoms will be assessed via modules. A score is generated for each dimension and standardized on a scale from 0 to 100, so that a high score reflects a high overall health status, a high functional level and a high symptomatic level. According to EORTC recommendations, the score can be calculated if at least 50% of the items in the corresponding dimension have been completed. Otherwise, the score will be considered missing.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-ELDerly 14 (QLQ-ELD14) | At enrolment, at 12 weeks, at 6 months and at 12 months
  The QLQ-ELD14 questionnaire is specific to elderly cancer patients. It contains 14 items measuring 7 dimensions of quality of life : two functional dimensions (maintaining a positive positive vision/motivation, family support) and 5 symptomatic dimensions (mobility, worries about others, worries about the future, disease burden, joint problems).
  All of the scales and single-item range in score from 0-100. A score is generated for each dimension, so that a high score reflects a high functional level (for the scales concerned), and a high symptomatic level (for the scales concerned).
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 13 (QLQ-LC13) | At enrolment, at 12 weeks, at 6 months and at 12 months
  The QLQ-LC13 is a lung cancer-specific questionnaire containing 13 items to assess symptoms specific to lung cancer and its treatment: dyspnea, cough, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, chest pain, arm or shoulder pain or shoulder pain, pain in other parts, anti-inflammatory drugs, drugs for pain. A score is generated per dimension so that a high score reflects a high symptomatic level.
  All of the scales and single-item range in score from 0-100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status represents a high quality of life, but a high score for symptom scale/item represents a high level of symptomatology/problems.
Geriatric characteristics G8 score | At enrollment and at disease progression for a maximum of 2-year-period.
  The following geriatric characteristics will be collected is available in the participant medical file: G8 score.
  The total G-8 score lies between 0 and 17. A higher score indicates a better health status.
Geriatric characteristics Geriatric Core DatasEt (G-CODE) | At enrollment and at disease progression for a maximum of 2-year-period.
  The following geriatric characteristics will be collected is available in the participant medical file: Geriatric Core DatasEt (G-CODE). G-CODE is a core set of geriatric data. It has ten tools/items and a median completion time of 9 min. It includes Katz autonomy scale (ADL), Instrumental Activities of Daily Living (IADL), Charlson score, mini Geriatric Depression Sale (mini-GDS), short cognitive impairment screening exam (mini COG), falls history, Timed Get Up and Go test, social environment.
  The G-CODE allows for a minimal geriatric description of the older cancer population and standardisation of geriatric data, enabling comparison across trials.

OTHER OUTCOMES:
Biobank sampling | At inclusion
  Blood samples will be collected at inclusion, before the first administration of NSCLC therapy, for exploratory analyses in ancillary studies

CONTACTS AND LOCATIONS:
Overall Officials: Laurent GREILLIER, Professor, Study Chair — Groupe Français de Pneumo-Cancérologie (GFPC)
Locations (41):
- France (41):
  - CH du Pays d Aix, Aix-en-Provence
  - Hôpital Henri Duffaut, Avignon
  - Institut du Cancer d'Avignon, Avignon
  - CH Bastia, Bastia
  - Oncologie Thoracique Hôpital Morvan, Brest
  - Pneumologie Centre François Baclesse, Caen
  - CH Métropole-Savoie, Chambéry
  - Centre Hospitalier du Cotentin, Cherbourg
  - CHU Hôpital Montpied, Clermont-Ferrand
  - Pneumologie Hospices Civils de Colmar, Colmar
  - Pneumologie CHI Creteil, Créteil
  - CH Elbeuf, Elbeuf
  - Polyclinique de Blois, La Chaussée-Saint-Victor
  - CHD Les Oudairies, La Roche-sur-Yon
  - CH La Rochelle, La Rochelle
  - Hôpital A. Mignot, Le Chesnay
  - Hôpital Robert Boulin, Libourne
  - CHU Dupuytren, Limoges
  - Hôpital de la Vallée - Service Pneumologie, Longjumeau
  - Centre Léon Bérard, Lyon
  - Hôpital Européen de Marseille, Marseille
  - Oncologie Thoracique Hôpital Nord, Marseille
  - GHEF Site de Meaux, Meaux
  - Centre d Oncologie de Gentilly, Nancy
  - Pneumologie CHR, Orléans
  - Pneumologie Hôpital Cochin, Paris
  - Pneumologie Hôpital Tenon, Paris
  - Cantre Catalan d Oncologie, Perpignan
  - CH Annecy Genevois, Pringy
  - Pneumologie CHI Quimper, Quimper
  - CHU Hôpital Ponchailloux, Rennes
  - Pneumologie Hôpital Charles Nicolle, Rouen
  - Pneumologie CHU Felix Guyon, Saint-Denis
  - Pneumologie CHU St Etienne, Saint-Etienne
  - Clinique Mutualiste, Saint-Nazaire
  - CHU de la Réunion, Saint-Pierre
  - CLCC Paul Strauss, Strasbourg
  - Hôpital d'Instruction des Armées Saint-Anne, Toulon
  - CHITS Toulon Sainte Musse, Toulon
  - Oncologie CHBA, Vannes
  - Hôpital Nord OUest, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: Undecided